CLINICAL TRIAL: NCT06300086
Title: Nationwide Utilization of Danish Government Electronic Letter System for Increasing Guideline-directed Medical Therapy in Chronic Kidney Disease
Acronym: NUDGE-CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: NUDGE-CKD
Record Dates: First submitted 2024-02-16; First posted 2024-03-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases; Behavior and Behavior Mechanisms
Keywords: Chronic Kidney Disease; Nudging; Behavioral Science; Guideline-directed medical therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Behavior

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient letters + no GP letter. (Experimental): Patients with CKD will receive digital nudge letters, but their associated GPs will not receive a digital nudge letter.
  The letters will inform patients with CKD of the importance of GDMT in CKD and that updated Danish guidelines for the treatment of CKD are available.
  Interventions: Behavioral: Electronically delivered nudging letters to patients with CKD
- Patient letters + GP letter. (Experimental): Patients with CKD and their associated GPs will receive digital nudge letters.
  The letters will inform the recipients of the importance of GDMT in CKD and that updated Danish guidelines for the treatment of CKD are available. The letter to the GPs will also include the definition of CKD and a summary of the guidelines.
  Interventions: Behavioral: Electronically delivered nudging letters to patients with CKD; Behavioral: Electronically delivered nudging letter to associated GPs of patients with CKD
- No patient letters + GP letter (Experimental): Patients with CKD will not receive digital nudge letters, but their associated GPs will receive a digital nudge letter.
  The letter will inform the GPs of the importance of GDMT in CKD and that updated Danish guidelines for the treatment of CKD are available. The letter will also include the definition of CKD and a summary of the guidelines.
  Interventions: Behavioral: Electronically delivered nudging letter to associated GPs of patients with CKD
- No patient letters + no GP letter (No Intervention): Neither patients with CKD nor their associated GPs will receive digital nudge letters.

INTERVENTIONS:
Behavioral: Electronically delivered nudging letters to patients with CKD — Patients in the active arm will receive a digital nudge letter as part of the study. The nudge letter will be delivered at baseline. Letters will be delivered through the official, mandatory Danish electronic letter system.
  The control arm will consist of patients with CKD randomized to not receive digital nudge letters (usual care).
  Other Names: Patient letters
  Arms: Patient letters + GP letter.; Patient letters + no GP letter.
Behavioral: Electronically delivered nudging letter to associated GPs of patients with CKD — The associated GPs of the patients in the active arm will receive one digital nudge letter as part of the study. The nudge letter will be delivered at baseline. The letters will be delivered through the official, mandatory Danish electronic letter system.
  The control arm will consist of patients with CKD whose associated GP was randomized to not receive a digital nudge letter (usual care).
  Other Names: GP letter
  Arms: No patient letters + GP letter; Patient letters + GP letter.

SUMMARY:
Kidney Disease Improving Global Outcomes (KDIGO) has recently updated the Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease (CKD). This update follows large placebo-controlled randomized trials, which established sodium-glucose cotransporter 2 inhibitors (SGLT2i) as an additional treatment option to reduce the risk of progression to kidney failure and cardiovascular disease in patients with CKD, both with and without diabetes or albuminuria. As a result, SGLT2i is now recommended to a broad range of CKD patients by KDIGO, along with established medical therapies such as renin-angiotensin system inhibition (RASi). Despite the significant adverse consequences of CKD and substantial evidence supporting guideline-directed medical therapy (GDMT) to improve patient outcomes, awareness of CKD among patients and providers remains disproportionately low. Innovative solutions are needed to increase awareness of CKD. Such a solution could potentially be the use of electronic nudge letters delivered to patients with CKD and their general practitioners (GPs) that highlight the importance of GDMT and inform them of updated guidelines.

This study will investigate whether digital nudge letters delivered via the official Danish electronic letter system directly to patients with CKD and their associated GPs will improve GDMT in patients with CKD when compared to no letters.

DETAILED DESCRIPTION:
The study is a prospective, 2x2 factorial, registry-based, randomized, open-label implementation trial. The study population will consist of Danish adults diagnosed with CKD. Participants will be identified through Danish nationwide health registries using codes from the International Classification of Diseases, 10th revision (ICD-10).

The primary objective of this study is to investigate the effects of electronically sent nudging letters delivered directly to (1) patients with CKD and, separately, (2) electronically sent nudge letters delivered to GPs of the included CKD patients on the primary outcome of use of GDMT defined as at least one prescription of RASi or SGLT2i 6 months after intervention delivery in patients with CKD.

Patients with CKD will be randomized (1:1) to either a control arm (no digital nudge letters sent to the patient) or an intervention arm (a digital nudge letter). GPs of the enrolled patients with CKD will be randomized (1:1) to a control arm (no digital nudge letters sent to the GP) or an intervention arm (a digital nudge letter). The letters will inform the recipients about the importance of GDMT in CKD and that updated Danish guidelines for treating CKD are available. The letter to the GPs will also include the definition of CKD and a summary of the guidelines.

The interventions will be delivered through the official, mandatory Danish electronic letter system. All subject data will be retrieved from the Danish nationwide registries except for information on intervention allocation. Endpoints will be retrieved at prespecified dates using prespecified search algorithms.

This study will coincide with the release of the updated clinical guidelines on the treatment of CKD by the Danish Society of Nephrology.

ELIGIBILITY:
Inclusion criteria

1. Age +18 years
2. Diagnosis of CKD defined as at least one hospital encounter with the following ICD-10 codes in the primary diagnostic positions within ≤ 5 years: N18- N19, I12, E102, E112, E132, E142.

Exclusion criteria

For patient-level intervention comparisons:

1) Exemption from the official, mandatory Danish electronic mailbox system.

For general practice-level intervention comparisons:

1. Individuals on a patient list of general practice clinics run by Danish administrative Regions.
2. Individuals not on a patient list of a general practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28388 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with any prescription of renin-angiotensin system inhibition and/or sodium-glucose cotransporter 2 inhibitors | within 6 months

SECONDARY OUTCOMES:
Number of participants with any prescription of renin-angiotensin system inhibition | within 6 months
Number of participants with any prescription of sodium-glucose cotransporter 2 inhibitors | within 6 months
Number of participants with a new prescription of renin-angiotensin system inhibition and/or sodium-glucose cotransporter 2 inhibitors | within 6 months
Number of participants with a new prescription of renin-angiotensin system inhibition | within 6 months
Number of participants with a new prescription of sodium-glucose cotransporter 2 inhibitors | within 6 months
Time from intervention delivery to a new prescription of renin-angiotensin system inhibition and/or sodium-glucose cotransporter 2 inhibitors | within 6 months
Time from intervention delivery to a new prescription of renin-angiotensin system inhibition | within 6 months
Time from intervention delivery to a new prescription of sodium-glucose cotransporter 2 inhibitors | within 6 months

OTHER OUTCOMES:
Number of participants with an increase in baseline daily RASi dosage | within 6 months
Number of participants with any prescription of mineralocorticoid receptor antagonists | within 6 months
Number of participants with any prescription of non-steroid mineralocorticoid receptor antagonists | within 6 months
Number of participants with any prescription of cholesterol-lowering medication | within 6 months
Number of participants with any prescription of glucagon-like peptide-1 analogue | within 6 months
Number of participants with any prescription of antidiabetic medication besides SGLT2i | within 6 months
Number of participants with any prescription of antidiabetic medication | within 6 months
Number of participants with any prescription of antihypertensive medication besides renin-angiotensin system inhibition | within 6 months
Number of participants with any prescription of antihypertensive medication | within 6 months
Number of participants with a new prescription of mineralocorticoid receptor antagonists | within 6 months
Number of participants with a new prescription of non-steroid mineralocorticoid receptor antagonists | within 6 months
Number of participants with a new prescription of cholesterol-lowering medication | within 6 months
Number of participants with a new prescription of glucagon-like peptide-1 analogue | within 6 months
Number of participants with a new prescription of antidiabetic medication besides sodium-glucose cotransporter 2 inhibitors | within 6 months
Number of participants with a new prescription of antidiabetic medication | within 6 months
Number of participants with a new prescription of antihypertensive medication besides renin-angiotensin system inhibition | within 6 months
Number of participants with a new prescription of antihypertensive medication | within 6 months
Change in number of antihypertensive medications | within 6 months
Number of participants referred to nephrology outpatient clinics | within 6 months
Number of participants with an assessment of urine albumine to creatine ratio | within 6 months
Number of participants with an assessment of plasma-creatinine. | within 6 months
Number of participants with an assessment of estimated glomerular filtration rate by creatinine | within 6 months
Number of participants with an assessment of hemoglobin A1c | within 6 months
Number of participants with an assessment of lipids | within 6 months
Number of participants recipient of influenza vaccination | within 6 months
Number of participants recipient of COVID-19 vaccination | within 6 months
Total number of visits to general practitioners | within 6 months
Time to first phone contact to a general practice | within 6 months
Time to first visit with a general practitioner | within 6 months
Number of participants with any prescription of renin-angiotensin system inhibition and/or sodium-glucose cotransporter 2 inhibitors | Within 1, 2, 5 and 10 years
Number of participants with any prescription of renin-angiotensin system inhibition | Within 1, 2, 5 and 10 years
Number of participants with any prescription of sodium-glucose cotransporter 2 inhibitors | Within 1, 2, 5 and 10 years
Number of participants with a new prescription of renin-angiotensin system inhibition and/or sodium-glucose cotransporter 2 inhibitors | Within 1, 2, 5 and 10 years
Number of participants with a new prescription of renin-angiotensin system inhibition | Within 1, 2, 5 and 10 years
Number of participants with a new prescription of sodium-glucose cotransporter 2 inhibitors | Within 1, 2, 5 and 10 years
Time from intervention delivery to prescription of renin-angiotensin system inhibition and/or sodium-glucose cotransporter 2 inhibitors | Within 1, 2, 5 and 10 years
Time from randomization to prescription of renin-angiotensin system inhibition | Within 1, 2, 5 and 10 years
Time from randomization to prescription of sodium-glucose cotransporter 2 inhibitors | Within 1, 2, 5 and 10 years
Number of participants who have discontinued renin-angiotensin system inhibition treatment. | Within 1, 2, 5 and 10 years
Number of participants who have discontinued sodium-glucose cotransporter 2 inhibition treatment. | Within 1, 2, 5 and 10 years
Rate of change in estimated glomerular filtration rate | Within 1, 2, 5 and 10 years
Rate of change in urine albumine to creatinine ratio | Within 1, 2, 5 and 10 years
Number of participants with any hospitalization | Within 1, 2, 5 and 10 years
Total number of all-cause hospitalizations | Within 1, 2, 5 and 10 years
All-cause mortality | Within 1, 2, 5 and 10 years
Number of participants with kidney failure defined as a composite of sustained estimated glomerular filtration rate <15ml/min/1.73m2, dialysis dependence and kidney transplantation | Within 1, 2, 5 and 10 years
Number of participants with kidney failure (alternative definition #1) defined as a composite of sustained estimated glomerular filtration rate <15ml/min/1.73m2, dialysis dependence, kidney transplantation and renal death | Within 1, 2, 5 and 10 years
Number of participants with kidney failure (alternative definition #2) defined as a composite of sustained estimated glomerular filtration rate <15ml/min/1.73m2, dialysis dependence, kidney transplantation, renal death, and cardiovascular death. | Within 1, 2, 5 and 10 years
Number of participants with acute dialysis | Within 1, 2, 5 and 10 years
Number of participants with acute kidney insufficiency | Within 1, 2, 5 and 10 years
Number of participants with incident heart failure, heart failure hospitalization, or cardiovascular death | Within 1, 2, 5 and 10 years
Number of participants with major adverse cardiovascular events defined as a composite of myocardial infarction, stroke, and cardiovascular death. | Within 1, 2, 5 and 10 years
Number of participants with major adverse cardiovascular events (alternative definition) defined as a composite of myocardial infarction, revascularization, stroke, and cardiovascular death. | Within 1, 2, 5 and 10 years
Number of participants with individual components of the renal/cardiovascular composite outcomes | Within 1, 2, 5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MSc, MPH, PhD, Principal Investigator — Study Principal Investigator Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.

REFERENCES:
- [Derived] Skaarup KG, Johansen ND, Brandi L, Lindhardt MK, Bech JN, Svensson M, Kristensen T, Thuesen AD, Knudsen MG, Kampmann JD, Hornum M, Orts B, Modin D, Lassen MCH, Janstrup KH, Claggett BL, Vaduganathan M, Bhatt AS, Van Spall HGC, Jensen JUS, Zannad F, Solomon SD, Moller A, Borg R, Birn H, Hansen D, Biering-Sorensen T. A Nationwide Factorial Randomized Trial of Electronic Nudges to Patients With Chronic Kidney Disease and Their General Practices for Increasing Guideline-Directed Medical Therapy: The NUDGE-CKD Trial. Circulation. 2025 Aug 12;152(6):369-383. doi: 10.1161/CIRCULATIONAHA.125.075403. Epub 2025 Jun 7. PMID 40481660
- [Derived] Skaarup KG, Johansen ND, Brandi L, Lindhardt MK, Bech JN, Svensson M, Kristensen T, Thuesen AD, Knudsen MG, Kampmann JD, Hornum M, Orts B, Modin D, Lassen MCH, Janstrup KH, Claggett BL, Vaduganathan M, Bhatt AS, Van Spall H, Jensen JUS, Zannad F, Solomon SD, Moller A, Borg R, Birn H, Hansen D, Biering-Sorensen T. Rationale and design of NUDGE-CKD: A nationwide randomized factorial trial of electronic nudges for increasing guideline-directed medical therapy in chronic kidney disease. Am Heart J. 2025 Sep;287:61-78. doi: 10.1016/j.ahj.2025.03.015. Epub 2025 Mar 31. PMID 40174694